CLINICAL TRIAL: NCT00349921
Title: Clonidine Versus Adenosine to Treat Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P01NS041386_TRIAL1; P01NS041386 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: pain; chronic pain; clonidine; adenosine; complex regional pain syndrome; CRPS; a2-adrenergic agonists; alpha2-adrenergic agonists
MeSH Terms: conditions — Pain; Chronic Pain; Complex Regional Pain Syndromes | interventions — Clonidine; Adenosine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- clonidine first, then adenosine (Active Comparator): clonidine given in first injection adenosine given in second injection
  Interventions: Drug: clonidine
- adenosine first, then clonidine (Active Comparator): adenosine given in first injection clonidine given in second injection
  Interventions: Drug: adenosine
- clonidine given first, then placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- adenosine given first, then placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clonidine — Clonidine-a drug commonly used to treat high blood pressure-has been shown to effectively treat neuropathic pain, is FDA-approved for administration via epidural (an injection given in the lower back), and is the third most commonly prescribed drug for chronic intrathecal (an injection into the cerebrospinal fluid) use in people with chronic pain.
  Other Names: duraclon
  Arms: clonidine first, then adenosine
Drug: adenosine — Adenosine-a drug commonly administered intravenously (into a vein) to treat certain types of abnormal heart rhythms-has been found to reduce areas of allodynia (pain caused by a stimulus that does not normally cause pain) after intrathecal, but not intravenous administration in people with neuropathic pain.
  Arms: adenosine first, then clonidine
Drug: placebo — inactive substance
  Other Names: dummy
  Arms: clonidine given first, then placebo
Drug: placebo — inactive substance
  Other Names: dummy
  Arms: adenosine given first, then placebo

SUMMARY:
The purpose of this study is to determine the effects of clonidine and adenosine on nerve pain.

DETAILED DESCRIPTION:
This study is part of a pain center grant that focuses on how pain, especially chronic neuropathic pain, alters the response to traditional and non-traditional analgesics (pain medications).

Clonidine-a drug commonly used to treat high blood pressure-has been shown to effectively treat neuropathic pain, is FDA-approved for administration via epidural (an injection given in the lower back), and is the third most commonly prescribed drug for chronic intrathecal (an injection into the cerebrospinal fluid) use in people with chronic pain.

Adenosine-a drug commonly administered intravenously (into a vein) to treat certain types of abnormal heart rhythms-has been found to reduce areas of allodynia (pain caused by a stimulus that does not normally cause pain) after intrathecal, but not intravenous administration in people with neuropathic pain.

Intrathecal clonidine relieves pain by actions on a2-adrenoceptors in the spinal cord, whereas adenosine relieves pain by actions on A1 adenosine receptors. Researchers believe that intrathecal adenosine and clonidine may prove to be excellent painkillers for nerve pain. Therefore, the goal of this study is to determine the effects of clonidine and adenosine on nerve pain.

After initial screening, baseline measurements, and training to learn to estimate pain accurately using thermal heat testing, a sample of spinal fluid will be taken from each participant. Participants then will be randomly chosen to receive either clonidine, adenosine, or placebo. After receiving the study medication, participants will be monitored, with their vital signs checked at 30, 60, 120, 180, and 240 minutes.

Duration of the study for participants is 2 weeks, and includes two visits to the research center, each lasting approximately 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex regional pain syndrome (CRPS), type I involving a lower extremity

Exclusion Criteria:

* Pregnancy
* Allergy to clonidine
* Currently taking clonidine or other direct a2-adrenergic agonists, or taking cholinesterase inhibitors
* Patients with any serious or unstable medical problems (heart, lung, liver, kidney, or nervous system disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences; Richard Rauck, M.D., Principal Investigator — The Center for Clinical Research
Locations (2):
- United States (2):
  - The Center for Clinical Research, 145 Kimel Park Drive, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Medical Center Boulevard, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 Subjects with chronic pain were recruited from the Center for Clinical Research. Each subject was scheduled for a study visit and randomized to receive spinal clonidine, spinal adenosine or placebo. The subject was scheduled for a second study visit and received the opposite treatment from the first visit.
Pre-assignment Details: 24 subjects consented and enrolled 2 subjects withdrawn prior to group assignment because they did not meet inclusion / exclusion criteria on second review
Groups:
- Clonidine First, Then Adenosine: Clonidine given during the first period and adenosine given during the second period
- Adenosine First, Then Clonidine: Adenosine given during the first period and adenosine given during the second
- Clonidine First, Then Placebo: Clonidine given as during the first period, then placebo during the second
- Adenosine First, Then Placebo: Adenosine given during the first period and placebo given during the second
Period: First Spinal Injection
Arm/Group | Clonidine First, Then Adenosine | Adenosine First, Then Clonidine | Clonidine First, Then Placebo | Adenosine First, Then Placebo
Started | 10 | 10 | 1 | 1
Completed | 9 | 10 | 0 | 1
Not Completed | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Second Spinal Injection
Arm/Group | Clonidine First, Then Adenosine | Adenosine First, Then Clonidine | Clonidine First, Then Placebo | Adenosine First, Then Placebo
Started | 9 (One patient experienced an adverse event after period one and did not participate in period two) | 10 | 0 | 1
Completed | 9 | 10 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adenosine Given First, Then Clonidine: adenosine given in first injection clonidine given in second injection
- Clonidine Given First, Then Placebo: clonidine given first placebo given in second injection
- Adenosine First, Then Placebo: adenosine given in first injection placebo given in second injection
- Total: Total of all reporting groups
Arm/Group | Clonidine First, Then Adenosine | Adenosine Given First, Then Clonidine | Clonidine Given First, Then Placebo | Adenosine First, Then Placebo | Total
Number analyzed (Participants) | 10 | 10 | 1 | 1 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 1 | 1 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (6.4) | 43.7 (10.8) | 19 (0) | 54 (0) | 43.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 1 | 1 | 14
  Male | 2 | 6 | 0 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 1 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number Meeting Success Criterion
Description: Verbal pain report 2 hours post injection compared to baseline verbal pain scores prior to injection
Time Frame: baseline and 2 hours
Population: The primary outcome measure will be % change in pain report 2 hr following injection, using a response criterion of 30% reduction in ongoing pain.
Measure: Number; unit: participants meeting success criterion
Groups:
- Clonidine: clonidine received as either first or second injection
- Adenosine: Adenosine received as either first or second injection
- Placebo: Placebo received as either first or second injection
Arm/Group | Clonidine | Adenosine | Placebo
Number analyzed (Participants) | 21 | 20 | 1
participants meeting success criterion | 10 | 5 | 0
Statistical Analysis 1: Comparison: Clonidine vs Adenosine; Null hypothesis is that there is no difference between the groups in proportion of patients meeting the success criterion of >30% reduction in visual analog scale pain 120 min after intrathecal injection; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Groups:
- Clonidine First, Then Placebo: clonidine given first placebo given in second injection
Arm/Group | Clonidine First, Then Adenosine | Adenosine First, Then Clonidine | Clonidine First, Then Placebo | Adenosine First, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No